CLINICAL TRIAL: NCT06586775
Title: Outcome of Complete Pulpotomy in Healthy and Type 2 Diabetic Patients in Permanent Teeth with Irreversible Pulpitis - a Preliminary Prospective Interventional Study.
Brief Title: Outcome of Complete Pulpotomy in Healthy and Type 2 Diabetic Patients in Permanent Teeth with Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Keerthana ENDO
Record Dates: First submitted 2023-12-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Irreversible Pulpitis; Diabetes Mellitus, Type 2; Healthy
Keywords: Pulpotomy; irreversible pulpitis; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pulpotomy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and the outcome assessor will be blinded with the participants preoperative characteristics and allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- diabetic group (Experimental): complete pulpotomy will be performed in teeth with irreversible pulpitis in diabetic patients.
  Interventions: Procedure: Pulpotomy
- Healthy group (Active Comparator): complete pulpotomy will be performed in teeth with irreversible pulpitis in systemically healthy patients.
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy — complete pulpotomy

SUMMARY:
Endodontic research on the effects of DM on pulp tissues is scarce. Diabetic human and animal histological research demonstrated a decreased reparatory response in the pulp, resulting in chronic pulp inflammation and reduced dentin bridge formation. To date, there is no human clinical trial examining the impact of diabetes mellitus on teeth with irreversible pulpitis. As a result of the paucity of data in the literature, there is a clinical dilemma whether to recommend vital pulp therapy techniques or root canal treatment in diabetic patients with irreversible pulpitis.

To the best of our knowledge, no prospective study has evaluated the outcome of complete pulpotomy in T2DM patients and healthy controls with irreversible pulpitis. The aim of this preliminary study is to compare and evaluate the success rates of pulpotomy in healthy and type 2 diabetes mellitus patients in mature permanent teeth presenting with clinical symptoms of irreversible pulpitis.

DETAILED DESCRIPTION:
Introduction:

Endodontic disease can affect both the pulp and the periapical areas of the tooth. The resultant immune-pathological reaction could be acute or chronic inflammation, depending on the ability of pulp and periapical tissue to respond to and recover from the noxious stimuli. T2DM has been recognized as a crucial factor affecting the pulpal and periapical tissues, in terms of susceptibility, progression, and healing. Endodontic research on the effects of DM on pulp tissues is scarce. Diabetic human and animal histological research demonstrated a decreased reparatory response in the pulp, resulting in chronic pulp inflammation and reduced dentin bridge formation. To date, there is no human clinical trial examining the impact of diabetes mellitus on teeth with irreversible pulpitis. As a result of the paucity of data in the literature, there is a clinical dilemma whether to recommend vital pulp therapy techniques or root canal treatment in diabetic patients with irreversible pulpitis.

To the best of our knowledge, no prospective study has evaluated the outcome of complete pulpotomy in T2DM patients and healthy controls with irreversible pulpitis. The aim of this preliminary study is to compare and evaluate the success rates of pulpotomy in healthy and type 2 diabetes mellitus patients in mature permanent teeth presenting with clinical symptoms of irreversible pulpitis.

AIM The aim of this study is to evaluate and compare the outcome of complete pulpotomy in healthy and type 2 diabetes mellitus patients presenting with clinical and radiographic signs and symptoms indicative of irreversible pulpitis.

OBJECTIVES

* To evaluate the clinical and radiographic success of pulpotomy with clinical and radiographic signs indicative of irreversible pulpitis.
* To investigate the effect of treatment outcome on glycated hemoglobin (HbA1c) in type 2 diabetic patients with irreversible pulpitis.

RESEARCH QUESTION Does the complete pulpotomy in type 2 diabetes mellitus patients is as effective as complete pulpotomy in healthy patients in mature permanent teeth presenting with clinical and radiographic signs and symptoms indicative of irreversible pulpitis? PICO

* P (Population) - Diabetic patients with mature permanent teeth with clinical and radiographic signs of irreversible pulpitis
* I (Intervention) - Complete pulpotomy in diabetic patients
* C (Comparison) - Complete pulpotomy in healthy patients
* O (Outcome) - Assessment of clinical and radiographic success at 3, 6 and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus with HbA1c > 6.5% with no other co-morbidities.
2. Age and gender matched healthy patients
3. Age between 18 - 70 years.
4. Mature permanent teeth with clinical and radiographic signs and symptoms indicative of irreversible pulpitis (PAI score ≤2)
5. Tooth showing positive response to pulp sensibility testing.

Exclusion Criteria:

1. Patients with immunocompromised diseases or systematic diseases (other than diabetes mellitus)
2. Smokers, pregnant and lactating women
3. Teeth with immature roots or retained deciduous tooth.
4. Bleeding could not be controlled in ≥8 minutes.
5. Tooth with signs and symptoms of apical periodontitis.
6. Tooth with probing depth more than 4mm.
7. Positive history of antibiotic use in the past 1 month or requiring antibiotic prophylaxis and/or analgesic usage in past 3 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender matched healthy control participants to the same gender diabetic individuals will be analyzed.
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Treatment outcome | 6 and 12 month follow-up.
  Outcome of complete pulpotomy in healthy and diabetic patients through clinical and radiographic findings.

SECONDARY OUTCOMES:
1) Effect of treatment on glycated haemoglobin levels in diabetic patients | 3 months post-treatment
  Changes in glycated haemoglobin levels

CONTACTS AND LOCATIONS:
Overall Officials: Dr.keerthana G, MDS, Principal Investigator — PGIDS
Locations (1):
- Dr.keerthana, Rohtak, Haryana, India